CLINICAL TRIAL: NCT00657748
Title: Evaluation of the Tolerance and Efficiency of a Combined Oral Therapy With Lithium and GTA in Patients With Canavan Disease
Brief Title: Lithium and Acetate for Canavan Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Leukodystrophy Association (Other)
Responsible Party: Yannick VACHER, Department Clinical Research and Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070803
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Canavan Disease; Infantile; Deficiency Disease; Aspartoacylase; Leukodystrophy, Spongiform
Keywords: Leukodystrophy; Canavan disease,; Aspartoacylase,; Lithium,; Glyceryl Triacetate
MeSH Terms: conditions — Canavan Disease; Deficiency Diseases | interventions — gluconic acid; Pharmaceutical Preparations; Triacetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lithium Gluconate (drug) Glyceryl Triacetate GTA (drug)

INTERVENTIONS:
Drug: Lithium Gluconate (drug) Glyceryl Triacetate GTA (drug) — Lithium 1.3 mEq/kg/day (three administrations a day)during the study GTA 500 mg/kg/day in four administrations a day during the study
  Other Names: Lithium Gluconate (drug); Glyceryl Triacetate, GTA (drug)

SUMMARY:
The aim of this study is to determine whether oral supplementation with lithium and acetate may improve the biological and clinical prognosis in patients with Canavan Disease.

DETAILED DESCRIPTION:
Canavan Disease is an autosomal recessive devastating demyelinating disease caused by a deficiency in Aspartoacylase (ASPA) enzyme. There is no available treatment. ASPA deficiency leads to:- the accumulation of high levels of N-acetylaspartate (NAA), involved in myelin degeneration and epilepsy;- the deficient synthesis of acetate in oligodendrocytes, that could impair CNS myelination.Lithium administration induces a decrease in NAA in the brain of the tremor rats (animal model for CD) and in one patient (JANSON, 2005). On the other hand, administration of acetate could improve myelination in Canavan patients.For this reason, we propose to combine both treatments: Lithium Gluconate and Glyceryl Triacetate (GTA). Eighteen patients, aged 1 to 15 years, will receive oral GTA or Lithium during 4 months, then both treatment in association during 6 months. Patients will be sequentially evaluated up to the end of the treatment and 2 months thereafter for:-tolerance of the therapy (careful monitoring of clinical and biological parameters).- efficacy of the therapy on clinical, biological and radiological parameters. Particularly, we will evaluate using MRI-spectroscopy and CSF samples the decrease in NAA and increase in acetate levels in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and biochemical diagnosis of Canavan disease

Exclusion Criteria:

* Renal disease
* Thyroid disease
* Cardiac disease
* Impossibility to perform brain MRI

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a decrease of the NAA peak (> 20%) or the appearance of an acetate peak at the end of the treatment (10 months), using spectroscopy-MRI. | 10 months

SECONDARY OUTCOMES:
Secondary outcomes will be assessed at 10 months (end of the treatment): -Improvement of neuromotor performances (GMFM and Mullen scales), spasticity, and neurological severity | 10 months
-Improvement of epilepsy (number of seizures) | 10 months
-Decrease in NAA and increase in acetate contents in fluids (CSF, plasma, urine). | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Aubourg, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Caroline Sevin, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

REFERENCES:
- [Result] Mathew R, Arun P, Madhavarao CN, Moffett JR, Namboodiri MA. Progress toward acetate supplementation therapy for Canavan disease: glyceryl triacetate administration increases acetate, but not N-acetylaspartate, levels in brain. J Pharmacol Exp Ther. 2005 Oct;315(1):297-303. doi: 10.1124/jpet.105.087536. Epub 2005 Jul 7. PMID 16002461
- [Result] Madhavarao CN, Arun P, Moffett JR, Szucs S, Surendran S, Matalon R, Garbern J, Hristova D, Johnson A, Jiang W, Namboodiri MA. Defective N-acetylaspartate catabolism reduces brain acetate levels and myelin lipid synthesis in Canavan's disease. Proc Natl Acad Sci U S A. 2005 Apr 5;102(14):5221-6. doi: 10.1073/pnas.0409184102. Epub 2005 Mar 22. PMID 15784740
- [Result] Janson CG, Assadi M, Francis J, Bilaniuk L, Shera D, Leone P. Lithium citrate for Canavan disease. Pediatr Neurol. 2005 Oct;33(4):235-43. doi: 10.1016/j.pediatrneurol.2005.04.015. PMID 16194720
- [Result] Baslow MH, Kitada K, Suckow RF, Hungund BL, Serikawa T. The effects of lithium chloride and other substances on levels of brain N-acetyl-L-aspartic acid in Canavan disease-like rats. Neurochem Res. 2002 May;27(5):403-6. doi: 10.1023/a:1015504031229. PMID 12064356
- See also: ELA (European Leukodystrophy Association) — http://www.ela-asso.com/